CLINICAL TRIAL: NCT00907842
Title: Prevention of Parastomal Hernias and Incisional Hernias in Old Stoma Wounds: a Pilot Study
Brief Title: Hernia Prevention in Stomas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marc Schreinemacher (Other)
Responsible Party: Sponsor-Investigator, Marc Schreinemacher, investigator, Academisch Ziekenhuis Maastricht
Organization: Academisch Ziekenhuis Maastricht (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: MEC09-2-052; NL27625.068.09
Record Dates: First submitted 2009-05-21; First posted 2009-05-25 (Estimated); Last update posted 2013-04-08 (Estimated); Status verified 2013-04

CONDITIONS: Incisional Hernia; Parastomal Hernia
Keywords: stoma
MeSH Terms: conditions — Incisional Hernia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- mesh placement (Experimental)
  Interventions: Device: Parietex Parastomal Mesh

INTERVENTIONS:
Device: Parietex Parastomal Mesh — mesh placed intraperitoneally around the stoma

SUMMARY:
Knowing that the risk of stoma associated herniation (parastomal or incisional) is 30-50% and the associated morbidity significant, standard placement of a prophylactic mesh upon stoma creation might prevent parastomal (or incisional herniation, after closure) and improve the quality of life of a large group of patients. This study is meant to be a pilot study to see whether the mesh related risks of infection and adhesion morbidity are acceptable if the mesh is placed intraperitoneally.

DETAILED DESCRIPTION:
The idea of a prophylactic mesh has been tested before in a Swedish randomized controlled trial (RCT) with the mesh placed upon end colostomy formation. Results suggest this procedure is the panacea against stoma associated herniations. The investigators still have unanswered questions however, about the size and ideal position of the mesh, possible complications (infection, adhesions) and the benefit in terms of quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with a life expectancy of at least one year
* Temporary stoma formation
* Signed informed consent
* Elective surgery
* Clean-contaminated abdomen

Exclusion Criteria:

* American Society of Anaesthesiologists (ASA) score IV or above
* Incapacitated adult or no signed informed consent
* Emergency procedure
* Contaminated or infected abdomen
* Residual intraperitoneal mesh
* Already injured part of the abdominal wall where the stoma will be sited
* Contraindication to laparoscopy
* Longterm use of corticosteroids and other immunosuppressive agents
* Current antibiotic therapy
* One of the following conditions: immune deficiency, chemotherapy, ascites, peritoneal dialysis, pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2010-04; Primary Completion 2013-02 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
postoperative complications after prophylactic mesh placement around a stoma (i.e., infection of the mesh and adhesions to the mesh) | one year after placement
incisional herniation at the old stoma wound | two years

SECONDARY OUTCOMES:
stoma complications (stenosis, bulging, prolapse, retraction, skin problems) | two years after placement

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Bouvy, MD, PhD, Study Director — Maastricht University Medical Centre; Marc Schreinemacher, MD, Principal Investigator — Maastricht University Medical Centre
Locations (1):
- Maastricht University Medical Centre, Maastricht, Netherlands

REFERENCES:
- [Background] Janes A, Cengiz Y, Israelsson LA. Preventing parastomal hernia with a prosthetic mesh: a 5-year follow-up of a randomized study. World J Surg. 2009 Jan;33(1):118-21; discussion 122-3. doi: 10.1007/s00268-008-9785-4. PMID 19011935
- [Background] Cingi A, Cakir T, Sever A, Aktan AO. Enterostomy site hernias: a clinical and computerized tomographic evaluation. Dis Colon Rectum. 2006 Oct;49(10):1559-63. doi: 10.1007/s10350-006-0681-4. PMID 17120189